CLINICAL TRIAL: NCT04687826
Title: Perioperative Fluid Therapy in Patients Undergoing Pancreaticoduodenectomy - How to Reduce Postoperative Complications
Brief Title: Perioperative Fluid Therapy in Patients Undergoing Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Piia Peltoniemi, M.D. Principal Investigator, Helsinki University Central Hospital
Other Study IDs: GDFT1517
Record Dates: First submitted 2020-12-20; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Complications
Keywords: pancreaticoduodenectomy; Clavien-Dindo classification; pancreatic fistulas
MeSH Terms: conditions — Postoperative Complications; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreaticoduodenectomy in 2015: Patients who underwent pancreaticoduodenectomy in 2015 got intraoperative fluid therapy in goal directed fluid therapy technique. Most of the patients spent the first postoperative night in ICU where the monitoring of urine output and fluid balance are more specific than in a normal ward.
  Interventions: Other: Goal directed fluid therapy
- Pancreaticoduodenectomy in 2017: Patients who underwent pancreaticoduodenectomy in 2017 got liberal intraoperative fluid therapy and most of the patients spent the first postoperative night in a regular ward.
  Interventions: Other: Liberal fluid therapy

INTERVENTIONS:
Other: Goal directed fluid therapy — Patients in 2015 got intraoperative fluid therapy in goal directed fluid therapy technique.
  Groups: Pancreaticoduodenectomy in 2015
Other: Liberal fluid therapy — Patients in 2017 got liberal intraoperative fluid therapy influenced by their anaesthesiologist.
  Groups: Pancreaticoduodenectomy in 2017

SUMMARY:
Postoperative complication rates in patients undergoing pancreaticoduodenectomy remain high although the operation techniques have developed a lot in recent years. There is evidence that restrictive intraoperative fluid therapy could decrease postoperative complication rates but the results of the former studies have been somewhat controversial. The aim of this study is to examine whether the intraoperative and postoperative fluid therapy affect to the postoperative complication rates in patients undergoing pancreaticoduodenectomy.

DETAILED DESCRIPTION:
The study is a retrospective cohort study. The first cohort consists of patients who underwent pancreaticoduodenectomy in year 2015 when intraoperative fluid therapy were managed using goal directed fluid therapy technique. The second cohort consists of patients who underwent pancreaticoduodenectomy in year 2017 when intraoperative fluid therapy were based on the consideration of the anaesthesiologist. In 2015 most of the patients spent the first postoperative night in the ICU where the fluid management and monitoring of the urine output and vital functions were more controlled than in the normal ward. In 2017 most of the patients got in the regular ward right after the surgery. The aim of the study is to examine whether there are differences in the amounts of the intraoperative and postoperative fluids between the cohorts and does the perioperative fluid therapy affect to the complication rates.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or over
* patients who underwent pancreaticoduodenectomy in 2015 or in 2017

Exclusion Criteria:

* patients whose patient record information is insufficient

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have underwent pancreaticoduodenectomy in years 2015 and 2017 are counted in the study.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Intraoperative fluid volume | The duration of the surgery
  The amount of fluid (crystalloids and albumin) patients got during the surgery
Postoperative complications (Clavien-Dindo classification) | Postoperative day 0-30
  The rate of severe Clavien-Dindo complications (3-5)

SECONDARY OUTCOMES:
Severe surgical complications | Postoperative day 0-30
  The rate of surgical complications (Clavien Dindo 3-5), without cardiopulmonary complications
Cardiopulmonary complications | Postoperative day 0-30
  The rate of cardiopulmonary complications e.g., congestive heart failure, pleural effusion, dyspnea.
Pancreatic fistulas | Postoperative day 0-30
  The rate of severe pancreatic fistulas (grade B-C)
Postoperative fluid volume | Postoperative day 0-3
  The amount of fluid patients got postoperatively
Intraoperative fluid balance | The duration of the surgery
  The change in intraoperative fluid intake (crystalloids, colloids, blood products) and fluid output (urine output, blood loss, evaporation) in millilitres and ml/kg.
Postoperative fluid balance | Postoperative day 1-3
  The change in postoperative fluid intake (crystalloids, colloids, blood products) and fluid output (urine output, secretion in drains etc.) in millilitres.

CONTACTS AND LOCATIONS:
Overall Officials: Piia Peltoniemi, M.D., Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No